CLINICAL TRIAL: NCT02366598
Title: Acute Food INtake Effect of Hemp Protein (A FINEH Protein) Trial - Part 1 - Acute Effects of Hemp Protein on Blood Glucose, Appetite, Blood Pressure and Food Intake.
Brief Title: A FINEH Protein Trial - Part 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Harvest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B2014:115
Record Dates: First submitted 2014-12-08; First posted 2015-02-19 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Prevention; Obesity Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 20g Hemp protein shake (Experimental): Hemp protein shake, 20 grams, given once at beginning of acute trial
  Interventions: Other: Hemp shake
- 40 g hemp protein shake (Experimental): Hemp protein shake, 40 grams, given once, at beginning of acute trial
  Interventions: Other: Hemp shake
- 20 g Soybean protein shake (Active Comparator): Soybean protein shake, 20 grams, given once, at beginning of acute trial
  Interventions: Other: Soybean shake
- 40 g Soybean protein shake (Experimental): Soybean protein shake, 40 grams, given once, at beginning of acute trial
  Interventions: Other: Soybean shake
- Control shake (Placebo Comparator): non-protein control shake, given once, at beginning of acute trial
  Interventions: Other: Control

INTERVENTIONS:
Other: Hemp shake — Hemp protein shake
  Arms: 20g Hemp protein shake; 40 g hemp protein shake
Other: Soybean shake — Soybean protein shake
  Arms: 20 g Soybean protein shake; 40 g Soybean protein shake
Other: Control — Non-protein shake
  Arms: Control shake

SUMMARY:
The objectives of this trial are to assess the health benefits of acute hemp protein consumption compared to soybean protein and a non-protein control on: 1) blood glucose, appetite and blood pressure for one hour following consumption, 2) food intake at an ad libitum meal one hour following consumption and 3) blood glucose, appetite and blood pressure following the ad libitum meal to determine the "second meal effect" of hemp protein.

ELIGIBILITY:
Inclusion Criteria:

* Normoglycemic (<5.6 mmol/L)
* Body mass index (BMI) of 18.5-29.9 kg/m2 Participants will be excluded if they regularly skip breakfast, smoke, or consuming medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year.

Exclusion Criteria:

* Restrained eaters
* Regularly skip breakfast
* Smokers
* Those who are active (organized activities or athletic training at a high intensity; ≥ 150 min per week of moderate to vigorous physical activity)
* Those on medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentration | 0-200 min
  Measured in blood by glucometer
Appetite | 0-200 min
  Measured by VAS Questionnaire
Food intake | 0-200 min
  Ad-libitum meal
Blood pressure | 0-200 min
  Measured by automated bood pressure cuff

SECONDARY OUTCOMES:
Palatability of treatments and meal | 5 -80 minutes
  Measured by VAS questionnaire
Physical comfort | 0 - 200 min
  Measured by VAS questionnaire
Energy/fatigue | 0 - 200 min
  Measured by VAS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods, Winnipeg, Manitoba, Canada